CLINICAL TRIAL: NCT06839612
Title: Evaluation of the Efficacy of the Two-point Method in Percutaneous Transhepatic Choledoscopy and the Influence of the Long-term Recurrence of Hepatolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shengyu Wang, MD, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z023121604
Record Dates: First submitted 2025-02-13; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hepatolithiasis; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two point method (Experimental)
  Interventions: Procedure: Two-point method
- Conventional PTCS (Active Comparator)
  Interventions: Procedure: Conventional PTCS

INTERVENTIONS:
Procedure: Two-point method — In the two-point method, the distal end of the drainage tube was passed over the duodenal and intestinal lumen of the common bile duct during PTCD operation. In the process of sinus dilation, guide wire was sent into the intestinal lumen through the drainage tube, and then the drainage tube was inserted into the intestinal lumen with the extract forceps under the duodenoscope in reverse order to drag the drainage tube into the intestinal lumen before being sent into the guide wire.Clamp the guide wire with the access pliers and slowly draw out the guide wire through the mouth. Expand the outer inlet skin.When the skin was 6mm, the epigastric PTCD tube was removed, the percutaneous nephrostomy dilator was placed through the guide wire, and the patient was instructed to be drawn by the assistant.The mouth end of the guide wire, the surgeon pulls the other end of the guide wire, so that the two ends of the guide wire fix in vitro to form a higher tension to Expand the skin.
  Arms: Two point method
Procedure: Conventional PTCS — PTCS can be divided into three steps: PTCD, sinus dilation, and lithotomy. In PTCD, we first performed intraoperative fluoroscopy, and punctured the biliary tract at a relatively straight Angle with the target biliary tract as far as possible. The distal end of the indenture drainage tube was inserted into the duodeno-intestinal cavity through the end of the common bile duct. The PTCD drainage tube was indwelled for 3-5 days.When the sinus was mature, we used dilated sheath tubes to dilate the sinus to 14-18Fr at a time, and used the working channel established by the choledochoscope to carry out net basket stone extraction. If large diameter stones were difficult to be extracted through the net basket, mechanical lithotomy was adopted to solve the problem, and conventional anti-inflammation was adopted in all patients after surgery. Cholangiography or epigastric CT were used to confirm complete removal of the stones after lithotomy.
  Arms: Conventional PTCS

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of the two-point approach in patients with intrahepatic bile duct stones。The main questions it aims to answer are:

① By comparing the technical success rate and clinical success rate of the two-point method and the non-two-point method, the clinical effect of the two methods was judged.

② To analyze the probability of short-term complications of the two-point method during the operation and to judge its safety.

③ Patients were followed up after the two-point method to determine the recurrence rate of stones and the probability of long-term complications.

The researchers will compare the two-point method with conventional PTCS to evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* PTCS were only used for the treatment of hepatolithiasis
* patients receiving PTCS for the first time.

Exclusion Criteria:

* PTCD failure and withdrawal from treatment due to patients' subjective wishes were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Technical success rate | up to 1 week
Clinical success rate | up to 1 week
Stone recurrence rate | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Bleeding | up to 2 weeks
Liver abscess | up to 2 weeks
Cholangitis | up to 2 weeks
Bile leakage | up to 2 weeks
Pancreatitis | up to 2 weeks
Thoracic complication | up to 2 weeks
Iatrogenic injury | up to 2 weeks